CLINICAL TRIAL: NCT03133637
Title: Effect of Ceftriaxone on Neonatal Jaundice
Brief Title: Ceftriaxone and Jaundice in Neonates
Acronym: CEFT
Status: Completed | Type: Observational
Sponsor: University of Rochester (Other)
Responsible Party: Sponsor
Other Study IDs: 29287
Record Dates: First submitted 2017-03-30; First posted 2017-04-28 (Actual); Last update posted 2021-04-06 (Actual); Status verified 2021-04

CONDITIONS: Jaundice and Sepsis in Neonates
MeSH Terms: conditions — Jaundice | interventions — Ceftriaxone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Ceftriaxone Arm
  Interventions: Drug: ceftriaxone

INTERVENTIONS:
Drug: ceftriaxone — Eligible infants will receive ceftriaxone as standard of care for sepsis

SUMMARY:
Ceftriaxone is an antibiotic often used for the management of sepsis. Neonates commonly have jaundice during the first postnatal week. Ceftriaxone will be given as standard of care for sepsis and investigators will observe the effect on jaundice.

ELIGIBILITY:
Inclusion Criteria:

* Term infants with sepsis requiring IV antibiotics for more than 3 days and who has total serum bilirubin 6-12 mg/dL and resolving by day 4 of life.

Exclusion Criteria:

* Infants with asphyxia (Apgar score <3 at 5 minutes), chromosomal disorder, failed hearing test at baseline, family history of hearing loss, unconjugated hyperbilirubinemia requiring phototherapy, TORCH infection, craniofacial malformations, listeria monocytogenes infection, and any clinical conditions which will preclude discharge to home.

Ages: 3 Days to 7 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Term neonates
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2016-03; Primary Completion 2019-08-31 (Actual); Study Completion 2019-08-31 (Actual)

PRIMARY OUTCOMES:
change in bilirubin binding assays | baseline and through study completion, an average of 1 hour

SECONDARY OUTCOMES:
Automated brain stem evoke response test | through study completion, an average of 1 hour

CONTACTS AND LOCATIONS:
Locations (1):
- University of Rochester Medical Center, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided